CLINICAL TRIAL: NCT02578381
Title: Boston Scientific COMET Wire Validation Study
Acronym: COMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: COMET
Record Dates: First submitted 2015-09-29; First posted 2015-10-19 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Stable Angina
Keywords: pressure wire; coronary angiogram; validation
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Boston Scientific PW versus St Jude PW (Experimental): Performance of Boston Scientific PW vs St Jude PW
  Interventions: Device: Boston Scientific Pressure Wire; Device: Validation of Boston Scientific pressure wire
- Boston Sci PW vs Boston Sci PW (Experimental): Boston Sci PW vs Boston Sci PW
  Interventions: Device: Boston Scientific Pressure Wire; Device: Validation of Boston Scientific pressure wire
- St Jude PW versus St Jude PW (Active Comparator): Performance of St Jude PW vs St Jude PW
  Interventions: Device: Validation of Boston Scientific pressure wire

INTERVENTIONS:
Device: Boston Scientific Pressure Wire — St Jude Medical Pressure Wire
  Arms: Boston Sci PW vs Boston Sci PW; Boston Scientific PW versus St Jude PW
Device: Validation of Boston Scientific pressure wire

SUMMARY:
Summary of Study Aims

To assess, in a randomised fashion:

1. performance of Boston Scientific Pressure Wire versus St Jude Pressure Wire
2. performance of Boston Scientific Pressure Wire versus Boston Scientific Pressure Wire
3. performance of St Jude Pressure Wire versus St Jude Pressure Wire

DETAILED DESCRIPTION:
Given the following key points of evidence, the optimal management of chest pain patients who come to diagnostic coronary angiography would more often be achieved if there was concomitant data with regard to the presence of patient-specific and lesion-specific ischaemia:

* that it is the presence and extent of reversible myocardial ischaemia (RMI) that dominates over coronary anatomy as a predictor of near term cardiovascular events, as well as symptom relief
* that prognostic benefit after revascularisation is greatest in patients with the largest pre-procedure ischaemic burden
* that intra-coronary pressure wire (PW) data are strongly correlated with subsequent cardiac events despite the binary nature of the test
* that stenting of coronary lesions that are PW negative has a worse outcome than optimal medical therapy (OMT)
* that PW-directed percutaneous coronary intervention (PCI) in multivessel disease is associated with a better clinical outcome than angiogram-directed PCI despite fewer treated lesions and less stents
* that PW-directed PCI improves prognosis compared to OMT
* that mismatch exists in up to 30-40% of lesions encountered at angiography between the visual appearance of the severity of the lesion and whether the lesion is "ischaemic" (and therefore a target for revascularisation) according to PW.

The availability of PW has been shown to have had a substantial effect on overall management of patients undergoing diagnostic coronary angiography (ie when options are still OMT/PCI and coronary artery bypass grafting (CABG) in several observation studies including RIPCORD and the French Registry.

Yet, despite the seemingly persuasive data summarised here, the uptake of PW at the diagnostic stage of the patient pathway is still low. There are, as yet, no suitably powered randomised trials using the PW systematically at the stage of diagnostic angiography and comparing outcome with management based upon angiography alone. This is the gap that will be filled by RIPCORD2.

RIPCORD2 will use the new Boston Scientific Pressure Wire (BSPW), which is currently undergoing first-in-man testing in Chile. The device has, of course, already been internally validated by Boston Scientific engineers and scientists, but the purpose of the COMET study is to provide independent and objective validation of the performance of BSPW using the performance of the St Jude Medical pressure wire (SJPW) as the reference, both using inter-wire and intra-wire measurements. Thus, not only will we assess the reproducibility of the measurements between the 2 wires, but the investigators will also compare reproducibility of measurements from 2 wires of the same manufacturer.

ELIGIBILITY:
Inclusion Criteria

* >18yrs age
* Written informed consent
* Patients scheduled for diagnostic angiography (and/or "standby" angiography)
* Clinical requirement for pressure wire assessment

Exclusion Criteria

* STEMI presentation
* Aorto-ostial disease
* Pregnancy
* CABG
* Contraindication to adenosine
* Creatinine >180umol/L
* Life threatening co-morbidity
* Severe valve disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Coronary artery pressure as measured by Boston Scientific Pressure Wire (BSPW) | Day one
  The study will involve the use of two pressure wires simultaneously in a coronary artery.
  The three randomisation groups will allow the comparison of pressure measurements between two different wires (BSPW vs SJPW) and will document consistency of readings within the same wire (BSPW vs BSPW or SJPW vs SJPW). Measurements will be undertaken using standard drug protocols. No additional drugs will be necessary for study purposes.
  * The first wire allocated at randomisation will be passed to the target measurement position in the artery
  * The second wire allocated at randomisation will be passed to exactly the same point in the vessel
  * Positioning of the wires will be confirmed by X-rays
  * Simultaneous measurements will be taken from the 2 pressure wires
  * If there is a narrowing in more than one vessel the process will be repeated for each vessel. Once the measurement has been taken, both wires will be removed.
Coronary artery pressure as measured by St Jude Medical Pressure Wire (SJPW) | Day one
  The study will involve the use of two pressure wires simultaneously in a coronary artery.
  The three randomisation groups will allow the comparison of pressure measurements between two different wires (BSPW vs SJPW) and will document consistency of readings within the same wire (BSPW vs BSPW or SJPW vs SJPW). Measurements will be undertaken using standard drug protocols. No additional drugs will be necessary for study purposes.
  * The first wire allocated at randomisation will be passed to the target measurement position in the artery
  * The second wire allocated at randomisation will be passed to exactly the same point in the vessel
  * Positioning of the wires will be confirmed by X-rays
  * Simultaneous measurements will be taken from the 2 pressure wires
  * If there is a narrowing in more than one vessel the process will be repeated for each vessel. Once the measurement has been taken, both wires will be removed.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Curzen, BM(Hons) PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Liverpool Heart & Chest NHS Foundation Trust, Liverpool, Merseyside
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No